CLINICAL TRIAL: NCT02708602
Title: Principal Investigator
Brief Title: Correlation Between the Polymorphism ofβ2 AR and the Labor Progress After Labor Analgesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Caijuan Li, Nanjing Maternity and Child Health Care Hospital, Nanjing Maternity and Child Health Care Hospital
Other Study IDs: NMCHC2016003
Record Dates: First submitted 2016-02-18; First posted 2016-03-15 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Labor Analgesia
Keywords: β2-adrenergic receptor; genetic polymorphisms; labor progress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (6):
- β2AR Arg16Arg (AA group): People with β2AR Arg16Arg genotype.
  Interventions: Genetic: β2AR polymorphism
- β2AR Arg16Gly (AG group): People with β2AR Arg16Gly genotype.
  Interventions: Genetic: β2AR polymorphism
- β2AR Gly16Gly (GG group): People with β2AR Gly16Gly genotype.
  Interventions: Genetic: β2AR polymorphism
- β2AR Gln27Gln (CC group): People with β2AR Gln16Gln genotype.
  Interventions: Genetic: β2AR polymorphism
- β2AR Gln27Glu (CG group): People with β2AR Gln27Glu genotype.
  Interventions: Genetic: β2AR polymorphism
- β2AR Glu27Glu (GG group): People with β2AR Glu27Glu genotype.
  Interventions: Genetic: β2AR polymorphism

INTERVENTIONS:
Genetic: β2AR polymorphism

SUMMARY:
Labor and delivery is a unique physiological experience of women. Inappropriate length of labor progress during vaginal delivery may produce great risks for mother and fetus. Especially the slow progress is one of the most important reasons for the occurrence of cesarean section during vaginal delivery, which still with a high incidence in recent years.Previous studies have found that there was a significant correlation between the genetic polymorphisms of β 2-adrenergic receptor (β2AR) and the duration of vaginal delivery.Therefore, the researchers intend to investigate the distribution of β2-adrenergic receptor (β2AR) genetic polymorphisms among Chinese parturient and observe the relationship between the genetic polymorphisms and labor process after labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Required labor analgesia
* Chinese
* Spontaneous labor

Exclusion Criteria:

* Contraindications for epidural analgesia
* Allergic to opioids and/or local anesthetics
* Failed to performing epidural catheterization
* Organic dysfunction
* Those who were not willing to or could not finish the whole study at any time
* Using or used in the past 14 days of the monoamine oxidase inhibitors
* Alcohol addictive or narcotic dependent patients
* Subjects with a nonvertex presentation or scheduled induction of labor
* Twin gestation and breech presentation

Ages: 23 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The parturient undergoing labor analgesia in our hospital. And the eligible parturient aged at 23-43, gestational age 35-42 weeks with an ASA grade I-II, who spontaneously choosing vaginal delivery mode with epidural analgesia.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
total labor process | up to about 24h
  time from the regular uterus contractions until completed childbirth, assessed up to about 24h
duration of the first stage | up to about 20h
  time from the regular uterus contractions to full cervix dilation,assessed up to about 20h
duration of the second stage | up to about 2h
  time from full cervix dilation to the complete childbirth, assessed up to about 2h
Maternal visual analogue scale | At time of initiation of analgesia and hourly thereafter until 2 hours postpartum (approximately 10 hours)
  At time of initiation of analgesia and hourly thereafter until 2 hours postpartum (approximately 10 hours)

SECONDARY OUTCOMES:
method of delivery | At time of placental delivery
  At time of placental delivery
Maternal modified Bromage scale | At time of initiation of analgesia and hourly thereafter until 2 hours postpartum (approximately 10 hours)
  At time of initiation of analgesia and hourly thereafter until 2 hours postpartum (approximately 10 hours)
Rescue boluses, n of rescue boluses, and the consumption of the ropivacaine/sufentanil mixture | At two hours postpartum
  At two hours postpartum
Maternal satisfaction with analgesia | At two hours postpartum
  At two hours postpartum
Use of oxytocin after analgesia | At twenty-four hours postpartum
  At twenty-four hours postpartum
Neonatal Apgar scale | At the first and fifth minutes after baby was born
  At the first and fifth minutes after baby was born
Maximal oxytocin dose | At twenty-four hours postpartum
  At twenty-four hours postpartum
Maternal heart rate, respiratory rate, and blood pressure | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
  At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
Neonatal weight | At delivery
  At delivery